CLINICAL TRIAL: NCT05865886
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Trial Evaluating Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of BI 1291583 One Tablet Once Daily Over 12 Weeks Versus Placebo in Adult Patients With Cystic Fibrosis Bronchiectasis (Clairafly™)
Brief Title: A Study to Test How Well BI 1291583 is Tolerated by People With Cystic Fibrosis Bronchiectasis (Clairafly™)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1397-0013; 2022-502835-21-00 (Registry Identifier: CTIS); U1111-1291-2567 (Registry Identifier: WHO Registry)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis; Bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 mg BI 1291583 (Experimental)
  Interventions: Drug: BI 1291583
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to BI 1291583

INTERVENTIONS:
Drug: BI 1291583 — Once daily oral administration of 5 milligram (mg) tablets of BI 1291583 for 12 weeks.
  Other Names: Verducatib
  Arms: 5 mg BI 1291583
Drug: Placebo to BI 1291583 — Once daily oral administration of tablets of placebo matching BI 1291583 for 12 weeks.
  Arms: Placebo

SUMMARY:
This study is open to adults aged 18 years and older with cystic fibrosis bronchiectasis.

The purpose of this study is to find out whether a medicine called BI 1291583 is tolerated by people with cystic fibrosis bronchiectasis. Participants are put randomly into 2 groups. One group takes BI 1291583 tablets and the other group takes placebo tablets. Placebo tablets look like BI 1291583 tablets but do not contain any medicine. Participants in both groups take 1 tablet once a day for 12 weeks. Participants have twice the chance of being placed in the BI 1291583 group than in the placebo group.

Participants are in the study for about 6 months. During this time, they visit the study site 7 times. At the visits, the doctors check the health of the participants and note any health problems that could have been caused by BI 1291583.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients when signing the informed consent ≥18 years
2. Historical clinical diagnosis of Cystic fibrosis (CF) (symptoms of CF and sweat chloride ≥ 60 mmol/L and/or 2 CF-causing Cystic fibrosis transmembrane conductance regulator (CFTR) mutations)
3. Investigator-confirmed diagnosis of Bronchiectasis (BE) by Computed tomography (CT) scan and clinical history consistent with BE (e.g., cough, chronic sputum production, recurrent respiratory infections). Subjects whose past chest CT records are not available will undergo a chest CT scan during Screening. Historical scans must not be older than 5 years
4. History of pulmonary exacerbations requiring antibiotic treatment. In the 12 months before Visit 1, patients must have had either:

   1. at least 2 exacerbations, or
   2. at least 1 exacerbation and an St. George's Respiratory Questionnaire (SGRQ) Symptoms score of >40 at screening visit 1 For patients on stable oral or inhaled antibiotics as chronic treatment for BE, at least one exacerbation must have occurred while on stable antibiotics.
5. Patients must be able to provide spontaneous or induced sputum samples. Further inclusion criteria apply.

Exclusion Criteria:

1. Moderate or severe liver disease (defined by Child-Pugh score B or C hepatic impairment) or Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) > 3.0x Upper limit of normal (ULN) at Visit 1
2. Estimated glomerular filtration rate (eGFR) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula < 30 mL/min at Visit 1
3. Absolute blood neutrophil count < 1,000/mm^3 (equivalent to < 1000 cells/μL or < 10^9 cells/L) at Visit 1
4. Any findings in the medical examination (including blood pressure (BP), pulse rate (PR), or electrocardiogram (ECG)) and/or laboratory value assessed at Visit 1 or during screening period that in the opinion of the investigator may put the patient at risk by participating in the trial
5. Positive serological tests for hepatitis B, hepatitis C (also confirmed with Hepatitis C virus ribonucleic acid (HCV RNA)), or human immunodeficiency virus (HIV) infection, or known infection status.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Northwell Health Physician Partners, New York, New York
- UZ Leuven, Leuven, Belgium
- Germany (4):
  - Charite Universitätsmedizin Berlin KöR, Berlin
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
- Italy (2):
  - Azienda Ospedaliera Meyer, Florence
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Netherlands (2):
  - Amsterdam UMC, location VUMC, Amsterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Hospital Universitari Vall D Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Badorrek P, Diefenbach C, Kogler H, Eleftheraki A, Seitz F, Hohlfeld JM. Novel cathepsin C inhibitor, BI 1291583, intended for treatment of bronchiectasis: Phase I characterization in healthy volunteers. Clin Transl Sci. 2024 Aug;17(8):e13891. doi: 10.1111/cts.13891. PMID 39175217
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blind, placebo-controlled, parallel group trial evaluating safety, tolerability, pharmacodynamics and pharmacokinetics of BI 1291583 one tablet once daily over 12 weeks versus placebo in adult patients with cystic fibrosis bronchiectasis (Clairafly™).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Participants with cystic fibrosis bronchiectasis administered orally once daily tablets of placebo matching BI 1291583 for 12 weeks.
- 5 mg BI 1291583: Participants with cystic fibrosis bronchiectasis administered orally once daily 5 milligram (mg) tablets of BI 1291583 for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | 5 mg BI 1291583
Started | 7 | 15
Completed (Completed planned treatment) | 7 | 14
Not Completed | 0 | 1
Not completed — Serious adverse event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): included all randomised patients who were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg BI 1291583 | Total
Number analyzed (Participants) | 7 | 15 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (9.4) | 32.3 (11.0) | 32.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 3 | 10 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 14 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 15 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Any Treatment Emergent Adverse Events
Description: Occurrence of any treatment emergent adverse events is expressed as percentages of participants with treatment emergent adverse events.
  Percentages are rounded to one decimal place.
Time Frame: From first dose of trial drug administration until last dose of trial drug administration plus 28 days of residual effect period, up to 16 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Groups:
- BI 1291583 5 mg: Participants with cystic fibrosis bronchiectasis administered orally once daily 5 milligram (mg) tablets of BI 1291583 for 12 weeks.
Arm/Group | Placebo | BI 1291583 5 mg
Number analyzed (Participants) | 7 | 15
Percentage of participants | 85.7 | 93.3

2. Secondary Outcome: Relative Change From Baseline in NE Activity, in Sputum, at Week 8 After First Drug Administration
Description: Relative change from baseline in neutrophil elastase (NE) activity, in sputum, at Week 8 after first drug administration is reported.
  Relative change from baseline at Week 8 in neutrophil elastase was calculated as below: Relative fluorescence unit (RFU) at Week 8-Relative fluorescence unit at baseline)*100%/Relative fluorescence unit at baseline.
Time Frame: Before the first drug administration (baseline: mean value of screening and Week 0 prior to the first treatment intake) and Week 8 after first study drug administration.
Population: Treated Set (TS): included all randomised patients who were documented to have taken at least one dose of investigational treatment. Only participants with a value at baseline and at Week 8 are reported.
Measure: Mean (Standard Deviation); unit: percent change in RFU
Arm/Group | Placebo | 5 mg BI 1291583
Number analyzed (Participants) | 7 | 13
percent change in RFU | 39.69 (134.67) | -65.95 (49.37)

3. Secondary Outcome: Area Under the Curve of BI 1291583 in Plasma Over a Uniform Dosing Interval Tau=6h After the First Dose (AUC0-6)
Description: Area under the curve of BI 1291583 in plasma over a uniform dosing interval tau=6h after the first dose (AUC0-6) is reported.
Time Frame: Before drug administration and 1 hour (h), 3.5h, 6h after administration of the first dose of BI 1291583 at Day 1.
Population: Pharmacokinetic set (PKS): This patient set included all patients from the treated set (TS) who provided at least one post-dose plasma BI 1291583 concentration that was not excluded due to a protocol deviation relevant to the evaluation of pharmacokinetic (PK), or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours *nanomole/Liter (h*nmol/L)
Arm/Group | 5 mg BI 1291583
Number analyzed (Participants) | 15
hours *nanomole/Liter (h*nmol/L) | 14.0 (65.3)

4. Secondary Outcome: Area Under the Curve of BI 1291583 in Plasma Over a Uniform Dosing Interval Tau=6h at Steady State (AUC0-6,ss)
Description: Area under the curve of BI 1291583 in plasma over a uniform dosing interval tau=6h at steady state (AUC0-6,ss) is reported.
Time Frame: Before drug administration at Day 85 and 1 hour (h), 3.5h, 6h after administration of BI 1291583 at Day 85.
Population: Pharmacokinetic set (PKS): This patient set included all patients from the treated set (TS) who provided at least one post-dose plasma BI 1291583 concentration that was not excluded due to a protocol deviation relevant to the evaluation of pharmacokinetic (PK), or due to PK non-evaluability. Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours *nanomole/Liter (h*nmol/L)
Arm/Group | 5 mg BI 1291583
Number analyzed (Participants) | 8
hours *nanomole/Liter (h*nmol/L) | 65.9 (64.5)

5. Secondary Outcome: Maximum Measured Concentration of BI 1291583 in Plasma After the First Dose
Description: Maximum measured concentration of BI 1291583 in plasma after the first dose is reported.
Time Frame: Before drug administration and 1 hour (h), 3.5h, 6h, and 8h after administration of the first dose of BI 1291583 at Day 1.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 5 mg BI 1291583
Number analyzed (Participants) | 15
nmol/L | 3.33 (74.4)

6. Secondary Outcome: Maximum Measured Concentration of BI 1291583 in Plasma at Steady State
Description: Maximum measured concentration of BI 1291583 in plasma at steady state is reported.
Time Frame: Before drug administration at Day 85 and 1 hour (h), 3.5h, 6h after administration of BI 1291583 at Day 85.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 5 mg BI 1291583
Number analyzed (Participants) | 14
nmol/L | 11.6 (69.9)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious Adverse Events and other adverse events: From first dose of trial drug administration until last dose of trial drug administration plus 28 days of residual effect period, up to 16 weeks.
Description: Treated Set (TS): included all randomised patients who were documented to have taken at least one dose of investigational treatment.
Arm/Group | Placebo | 5 mg BI 1291583
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/7 | 5/15
Other Adverse Events (participants affected / at risk) | 6/7 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | 5 mg BI 1291583 (N=15)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 3
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | 5 mg BI 1291583 (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 1
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 0 | 2
Otitis externa (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Sputum purulent (Infections and infestations) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Forced expiratory volume decreased (Investigations) | 0 | 2
Prothrombin time prolonged (Investigations) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Hypotonia (Nervous system disorders) | 0 | 1
Sleep deficit (Nervous system disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT05865886/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT05865886/SAP_001.pdf